CLINICAL TRIAL: NCT02444533
Title: A Phase IV Randomize, Single-Blind, Trial of Liposomal Bupivacaine (EXPAREL®) for Pain Control in Post-Tonsillectomy Patients
Brief Title: EXPAREL® for Pain After Tonsillectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Daniel L. Price, M.D., PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-007071
Record Dates: First submitted 2015-05-08; First posted 2015-05-14 (Estimated); Results first posted 2017-07-14 (Actual); Last update posted 2017-07-14 (Actual); Status verified 2017-06

CONDITIONS: Tonsillectomy; Tonsillitis; Post-operative Pain
Keywords: Liposomal Bupivacaine
MeSH Terms: conditions — Tonsillitis; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Liposomal Bupivacaine (Active Comparator): Patient will receive liposomal bupivacaine in the tonsillar fossae after tonsillectomy
  Interventions: Drug: Liposomal Bupivacaine
- No treatment (No Intervention): Patient will not be given any medications in the tonsillar fossae after tonsillectomy

INTERVENTIONS:
Drug: Liposomal Bupivacaine — Injection of 8 ml of liposomal bupivacaine total in the tonsillar fossae after tonsillectomy.
  Other Names: Exparel
  Arms: Liposomal Bupivacaine

SUMMARY:
The purpose of this study is to determine whether liposomal bupivacaine (long acting injectable anesthetic) provides greater post operative pain relief compared to the standard post operative pain regiment for tonsillectomy patients.

DETAILED DESCRIPTION:
Subjects will be screened in the clinic when being evaluated for indications for tonsillectomy. Once the decision to proceed with tonsillectomy is made, the patient will be given the information on the study, provided time to review the information and interested patients will be consented.

There will be two stages in the study. The first will be the operative stage, which includes the injection during the operation. The second stage is the patient participation stage. During this stage, the patient records the amount of oral pain medication usage, oral intake after their procedure, in addition to their pain scores. These scores are recorded and brought back (or mailed in) to the clinic for collection during the follow up visit, approximately 1 month later (patients will keep records for two weeks). The patients will be freed from participation in the study after the one month visit.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of recurrent tonsillitis or bilateral tonsillar hypertrophy requiring bilateral tonsillectomy
* Willing and able to understand and provide written informed consent

Exclusion Criteria:

* Known pregnancy
* Women who are currently nursing a child
* History of coagulopathy; such as hemophilia or Von Willebrand disease, or any congenital or acquired bleeding disorder
* Use of anticoagulation medication during the study, i.e. aspirin, Coumadin, Plavix, or medications similar in class to these medications will exclude the patient from participation
* Inability to provide informed consent (patients under guardianship)
* Known hypersensitivity to local anesthetics
* History of cardiac disease; such as current impaired cardiovascular function, past history of myocardial infarction, congenital heart disease, current cardiac symptoms, i.e. angina, shortness of breath, or chest pain as determined by history or review of the medical record.
* History of complex pulmonary disease; such as uncontrolled asthma, chronic obstructive pulmonary disease (COPD), or interstitial lung disease as determined by history or review of the medical record.
* Impaired renal function as documented in the medical record in the last 3 months with a serum creatinine greater than 1.2 mg/dL or glomerular filtration rate < 60 mL/min/body surface area (BSA) as determined by history or review of the medical record.
* History of or current hepatic disease as documented by liver function test abnormality in the last 3 months as determined by history or review of the medical record.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2015-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel L Price, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at the Mayo Clinic in Rochester, Minnesota.
Period: Overall Study
Arm/Group | Liposomal Bupivacaine | No Treatment
Started | 17 | 22
Completed | 15 | 18
Not Completed | 2 | 4
Not completed — Not able to complete forms | 0 | 2
Not completed — Only gave post-procedure complications | 2 | 2

BASELINE CHARACTERISTICS:
Population: Demographics include only subjects who were reported as having at least partial outcome data.
Groups:
- Total: Total of all reporting groups
Arm/Group | Liposomal Bupivacaine | No Treatment | Total
Number analyzed (Participants) | 15 | 18 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 18 | 33
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 15 | 23
  Male | 7 | 3 | 10
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 18 | 33

OUTCOME MEASURES:

1. Primary Outcome: Pain Score (Pain Scores on a 0/10 Scale)
Description: Subjects recorded pain scores four times a day in a daily pain diary using a Visual Analog Scale with markings from 0 to 10. 0 indicated "no pain" and 10 indicated "worst possible pain"
Time Frame: day of surgery, 14 days after surgery
Population: Results include only subjects who were reported as having at least partial outcome data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Liposomal Bupivacaine | No Treatment
Number analyzed (Participants) | 15 | 18
units on a scale
  day of surgery | 3.07 (2.03) | 4.9 (2.79)
  14 days after surgery | 1.76 (1.44) | 1.42 (1.04)
Statistical Analysis 1: Comparison: Liposomal Bupivacaine vs No Treatment; Comparison between groups for pain on day of surgery. Statistical significance was defined as a p-value less than 0.05; Test type: Superiority; p = 0.043, t-test, 2 sided
Statistical Analysis 2: Comparison: Liposomal Bupivacaine vs No Treatment; Comparison between groups for pain at 14 days after surgery. Statistical significance was defined as a p-value less than 0.05; Test type: Superiority; p = 0.445, t-test, 2 sided

2. Primary Outcome: Pain Medication Usage (Milligrams Used)
Description: Subjects recorded pain medication usage in milligrams used of Tylenol, Ibuprofen, and Oxycodone over a 2 week time frame
Time Frame: 2 weeks after surgery
Population: One subject on the no treatment arm was excluded for lack of follow up data, therefore 18 (from participant flow) -1 = 17.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Liposomal Bupivacaine | No Treatment
Number analyzed (Participants) | 15 | 17
mg
  Ibuprofen (Motrin) | 14013 (18109) | 9753 (11509)
  Acetaminophen (Tylenol) | 30615 (13196) | 31287 (13185)
  Oxycodone (OxyContin) | 265 (246) | 244 (159)
Statistical Analysis 1: Comparison: Liposomal Bupivacaine vs No Treatment; Comparison between groups for ibuprofen usage. Statistical significance was defined as a p-value less than 0.05; Test type: Superiority; p = 0.650, t-test, 2 sided
Statistical Analysis 2: Comparison: Liposomal Bupivacaine vs No Treatment; Comparison between groups for acetaminophen usage. Statistical significance was defined as a p-value less than 0.05; Test type: Superiority; p = 0.970, t-test, 2 sided
Statistical Analysis 3: Comparison: Liposomal Bupivacaine vs No Treatment; Comparison between groups for oxycodone usage. Statistical significance was defined as a p-value less than 0.05; Test type: Superiority; p = 0.835, t-test, 2 sided

3. Primary Outcome: Oral Intake (Patient Recorded Oral Intake)
Description: Subjects recorded oral intake over one week after surgery
Time Frame: 1 week after surgery
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Liposomal Bupivacaine | No Treatment
Number analyzed (Participants) | 15 | 18
mL | 13715 (7551) | 12492 (4271)
Statistical Analysis 1: Comparison: Liposomal Bupivacaine vs No Treatment; Comparison between groups at 7 days. Statistical significance was defined as a p-value less than 0.05; Test type: Superiority; p = 1.0, t-test, 2 sided

4. Secondary Outcome: Number of Subjects Experiencing Complications ( Allergic Reaction, Swallowing Dysfunction, Hospital Admission Related to the Study Drug)
Description: Patients will be monitored for drug related complications such as allergic reaction, swallowing dysfunction, hospital admission related to the study drug.
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Liposomal Bupivacaine | No Treatment
Number analyzed (Participants) | 15 | 18
Participants
  Allergic reaction | 0 | 0
  Swallowing dysfunction | 0 | 0
  Hospital admission related to the study drug | 0 | 0

5. Secondary Outcome: Number of Subjects With Post-tonsillectomy Bleeding
Description: The rate of post-tonsillectomy bleeding will be recorded and compared to the arm who did not receive the injection.
Time Frame: 4 weeks
Population: In the Liposomal Bupivacaine arm, 15 subjects had data on the primary endpoints, and an additional 2 provided information regarding post-procedure complications, but didn't provide data on other outcomes, therefore the analysis population for the Liposomal Bupivacaine is 17.
Measure: Count of Participants; unit: Participants
Arm/Group | Liposomal Bupivacaine | No Treatment
Number analyzed (Participants) | 17 | 18
Participants
  Any form of bleeding | 4 | 2
  Required a trip back to the operating room | 2 | 1
  No bleeding | 11 | 15

ADVERSE EVENTS:
Time Frame: 5 weeks post surgery
Arm/Group | Liposomal Bupivacaine | No Treatment
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/22
Other Adverse Events (participants affected / at risk) | 0/17 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes